CLINICAL TRIAL: NCT01728090
Title: Effectiveness of a Handwashing Programme in the Prevention of School Absenteeism Due to Respiratory Infections
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación Pública Andaluza para la Investigación Biomédica Andalucía Oriental (Other)
Collaborators: Ministry of Health, Spain (Other Government)
Responsible Party: Principal Investigator, Ernestina Azor Martínez, MD, PhD, Fundación Pública Andaluza para la Investigación Biomédica Andalucía Oriental
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PI 0388/2008
Record Dates: First submitted 2012-11-13; First posted 2012-11-16 (Estimated); Last update posted 2012-11-19 (Estimated); Status verified 2012-11

CONDITIONS: Upper Respiratory Infections; Influenza; Common Cold
Keywords: handwashing; hand sanitizer; absenteeism; school age children; preschool children
MeSH Terms: conditions — Respiratory Tract Infections; Influenza, Human; Common Cold | interventions — Hand Sanitizers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hand sanitizer (Experimental): Intervention classrooms received alcohol-based hand sanitizer and a programme educational.
  Characteristics of the hydroalcoholic gel (ALCO ALOE GEL): chlorhexidine digluconate at 20% solution, phenoxyethanol 1%, benzalkonium chloride 0.%. aloe Barbadensis 5%, Renat ethyl alcohol 70%, excipients c.s.p. 100 ml. Alcohol of between 65 - 70% degrees, pondus Hydrogenium (pH) = 7-7,5.
  Interventions: Other: hand sanitizer
- Control (No Intervention): No hand sanitizer or educational programme were used

INTERVENTIONS:
Other: hand sanitizer — alcohol-based, hydroalcoholic gel
  Other Names: ALCO ALOE GEL
  Arms: Hand sanitizer

SUMMARY:
The aim of the study was to assess the effectiveness of a hand-washing programme using hand sanitizer in the prevention of school absenteeism due to upper respiratory infections. Students in intervention classrooms used hand sanitizers at schools and a programme educational on hand hygiene. The investigators hypothesize that the use de hand sanitizers in elementary school will reduce absenteeism due to upper respiratory infections.

DETAILED DESCRIPTION:
School absenteeism due to respiratory infections is one of the greatest problems in schools. Its high incidence and easy transmission among pupils have a great impact requiring a vast number of medical visits, hospitalisations, use of antibiotic and antipyretic treatments, symptomatic medication, etc. besides being a cause for school absenteeism and time off work for parents. Hand- washing is the most important and effective measure to prevent the transmission of infections. The investigators evaluated the effectiveness of a hand-washing programme using hand sanitizer in the prevention of school absenteeism due to upper respiratory infections.

A cluster randomised, controlled and open study of 2 cohorts of primary school children between the ages of 4 and 12, attending 5 Public Schools in a geographic area of the Almería province (Spain). This study was carried out throughout the 8 months of an academic year (October 2009 to May 2010). The experimental group washed their hands with soap and water, complemented with hand sanitizer, while the control group followed usual hand washing. The parents of both groups completed the survey on sociodemographic characteristics and questions about hand hygiene referred to when and how their children wash their hands Progenitors of children who were absent from school collected upper respiratory infections symptoms and handed in the completed form to the teacher. One Research assistant collected the absence sheets of the participating classes weekly, telephoned the parents of absent children to enquire about the cause of their absence, visited the classrooms and collaborated with the teachers in hand hygiene related activities.

ELIGIBILITY:
Inclusion criteria:

* School children between the ages of 4 and 12 years old, enrolled in the above mentioned public schools,
* The parents/tutors signed an agreement after being informed of its content.

Exclusion criteria:

* Children with absenteeism due to a different cause from upper respiratory infections
* Children with chronic illnesses that could affect their likelihood of contracting an infection or the duration of their period of absence from school
* Children whose parents did not authorise their participation in the study.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1640 (Actual)
Dates: Start 2009-10; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
School absenteeism rate caused by upper respiratory infection | One academic year (eight months follow-up)
  The incidence rate of respiratory infections was calculated dividing the number of episodes respiratory by the number of pupils during the period of this study who were susceptible to the infection.
  Incidence rate ratio indicates (IRR): the ratio between incidence rate in both study groups.

SECONDARY OUTCOMES:
Average duration of absence | One academic year (eight months follow-up)
  The average duration of absence per child was calculated dividing the number of absence days due to respiratory infection by the total number of children during that period.

CONTACTS AND LOCATIONS:
Overall Officials: Ernestina Azor, MD, PhD, Principal Investigator — Department of Health of Andalusia